CLINICAL TRIAL: NCT03508466
Title: Investigation of the Underlying Mechanism of Hypersensitivity Reactions to Intravenous Iron Nanomedicines in Patients With Previous Hypersensitivity Reaction Compared to Controls - a Cross-sectional Study
Brief Title: Mechanism of Hypersensitivity Reactions to Iron Nanomedicines
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01606; sp18Steveling (Other: CTU)
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Iron-deficiency
Keywords: hypersensitivity
MeSH Terms: conditions — Anemia, Iron-Deficiency; Hypersensitivity | interventions — Sensitivity and Specificity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: adult participants from 18-65 years of age previous hypersensitivity reaction grades I-IV to intravenous ferric carboxymaltose (Ferinject)
  Interventions: Behavioral: hypersensitivity reaction
- Group 2: adult participants from 18-65 years of age previous intravenous ferric carboxymaltose (Ferinject) and no hypersensitivity reaction
- Group 3: adult participants from 18-65 years of age previous hypersensitivity reaction grades I-IV to iron sucrose (Venofer)
  Interventions: Behavioral: hypersensitivity reaction
- Group 4: adult participants from 18-65 years of age previous intravenous iron sucrose (Venofer) and no hypersensitivity reaction

INTERVENTIONS:
Behavioral: hypersensitivity reaction — Previous hypersensitivity reaction
  Groups: Group 1; Group 3

SUMMARY:
Iron deficiency is common and when oral treatment is not sufficient intravenous application is indicated. Hypersensitivity to intravenous iron nanomedicines is rare but does occur and little is known about the underlying mechanism but complement activation has been suggested.

This is a purely exploratory study as it is not yet known whether in vitro complement activation can be stimulated by titration with iron preparations. These data will provide first empirical evidence of whether and to what extent complement activation occurs in this population.

ELIGIBILITY:
Inclusion Criteria:Group 1)

* adult participants from 18-65 years of age
* previous hypersensitivity reaction grades I-IV to intravenous ferric carboxymaltose (Ferinject) Group 2)
* adult participants from 18-65 years of age
* previous intravenous ferric carboxymaltose (Ferinject) and no hypersensitivity reaction Group 3)
* adult participants from 18-65 years of age
* previous hypersensitivity reaction grades I-IV to iron sucrose (Venofer) Group 4)
* adult participants from 18-65 years of age
* previous intravenous iron sucrose (Venofer) and no hypersensitivity reaction

Exclusion Criteria:

* Group 1)-4) • Autoimmune disorder or immune deficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants with a previous hypersensitivity reaction to an iron nanomedicine application and participants without a hypersensitivity reaction to a previous iron nanomedicine application
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Complement activation | At baseline
  The primary outcome, complement activation, will be measured by the respective concentrations of the complement compounds sC5b9, C4d, C3a and C5a (ng/ml), and CP, LP and AP (%) 30 minutes after titration of two concentrations (100 ng/ml and 500 ng/ml) of Ferinject and Venofer into serum probes. That is for each subject, four serum probes will be analysed (100 ng/ml Ferinject, 500 ng/ml Ferinject, 100 ng/ml Venofer and 500 ng/ml Venofer).

CONTACTS AND LOCATIONS:
Overall Officials: Esther H Steveling-Klein, Dr., MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland